CLINICAL TRIAL: NCT02967159
Title: A RANDOMIZED OPEN LABEL CROSS-OVER STUDY TO EVALUATE PHARMACOKINETICS AND SAFETY OF SINGLE INHALED DOSES OF ABEDITEROL AND AZD7594 GIVEN ALONE, IN FIXED DOSE COMBINATION (FDC) AND IN FREE COMBINATION, USING DPI, IN MALE HEALTHY VOLUNTEERS
Brief Title: A Study to Evaluate the Disposition of Drug in Body and Safety After Administration of Single Inhaled Doses of Drugs Abediterol and AZD7594 Administered Alone, in Fixed Dose Combination and in Free Combination Using the Dry Powder Inhaler in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D7110C00001
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma
Keywords: chronic obstructive pulmonary disease (COPD); asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — 5-(2-((6-(2,2-difluoro-2-phenylethoxy)hexyl)amino)-1-hydroxyethyl)-8-hydroxyquinolin-2(1H)-one; velsecorat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Abediterol ) (Experimental): Treatment A: The subjects will receive Abediterol 2.5 μg via DPI
  Interventions: Drug: Abediterol
- Treatment B (AZD7594) (Experimental): Treatment B: The subjects will receive AZD7594 440 μg via DPI
  Interventions: Drug: AZD7594
- Treatment C (AZD7594/abediterol ) (Experimental): Treatment C: The subjects will receive AZD7594/ abediterol 440 μg/2.5 μg FDC via DPI
  Interventions: Drug: AZD7594/abediterol
- Treatment D (AZD7594 and abediterol) (Experimental): Treatment D: The subjects will receive AZD7594 440 μg and abediterol 2.5 μg free combination administered via 2 separate DPIs
  Interventions: Drug: AZD7594 and abediterol

INTERVENTIONS:
Drug: Abediterol — Treatment A: Abediterol 2.5 μg via DPI
  Other Names: Treatment A
  Arms: Treatment A (Abediterol )
Drug: AZD7594 — Treatment B: AZD7594 440 μg via DPI
  Other Names: Treatment B
  Arms: Treatment B (AZD7594)
Drug: AZD7594/abediterol — Treatment C: AZD7594/abediterol 440 μg/2.5 μg FDC via DPI
  Other Names: Treatment C
  Arms: Treatment C (AZD7594/abediterol )
Drug: AZD7594 and abediterol — Treatment D: AZD7594 440 μg and abediterol 2.5 μg free combination administered via 2 separate DPIs
  Other Names: Treatment D
  Arms: Treatment D (AZD7594 and abediterol)

SUMMARY:
AZD7594 is a non steroidal, potent and selective modulator of the glucocorticoid receptor (GR) under development for once daily inhaled treatment of chronic obstructive pulmonary disease (COPD) and asthma. Abediterol is a novel and selective β2 adrenergic receptor agonist with the potential for once daily treatment of asthma and COPD in fixed dose combination (FDC) with an ICS or a novel anti inflammatory (AI) agent. This study will be the first clinical study for the combination exposure of AZD7594 with abediterol as 2 compounds in FDC or in free combination via 2 separate dry powder inhalers (DPIs). This study will be conducted in healthy male subjects to minimize the effects of concomitant disease states or medications on study measurements.

DETAILED DESCRIPTION:
AZD7594 is a non steroidal, potent and selective modulator of the glucocorticoid receptor (GR) under development for once daily inhaled treatment of chronic obstructive pulmonary disease (COPD) and asthma. Inhaled corticosteroids (ICS) have not been definitively shown to decrease the rate of decline in lung function that is typical of COPD. The aim is to develop AZD7594 as a well tolerated once daily selective inhaled GR modulator with an acceptable side effect profile compared to conventional ICS on the market. Abediterol is a novel and selective β2 adrenergic receptor agonist with the potential for once daily treatment of asthma and COPD in fixed dose combination (FDC) with an ICS or a novel anti inflammatory (AI) agent Fixed dose ICS/LABA combination treatment is more effective in improving lung function, health status and reducing exacerbations than the individual components. The long term goal of abediterol development program in COPD is to investigate it both as a monotherapy and as a combination therapy in conjunction with an ICS or a novel anti inflammatory agent. This study will be the first clinical study for the combination exposure of AZD7594 with abediterol as 2 compounds in FDC or in free combination via 2 separate dry powder inhalers (DPIs). This study will be conducted in healthy male subjects to minimize the effects of concomitant disease states or medications on study measurements. Subjects will receive all 4 treatments in a randomized order. Given that the treatment in each period is a single dose of AZD7594, a 21 (±2) day wash out should be adequate to prevent carry over effect to next period. The abediterol elimination half life is shorter than that of AZD7594. Therefore, a 21 (±2) day wash out is sufficient for the elimination of both AZD7594 and abediterol. Overall, pre-clinical and clinical data generated to date with abediterol show expected safety profile, and support the continued studies with abediterol.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male subjects aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture
3. Have a body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Subjects should be willing to follow reproductive restrictions #11 in Section 7.47.4.1 to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm or fathering a child from the first day of dosing until 3 months after the last dose of IMP.
5. Be able to inhale from the DPI devices according to given instructions.
6. Able to understand, read and speak the German language.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Known Gilbert's syndrome, family history of Gilbert's syndrome or suspicion of Gilbert's syndrome based on liver function tests.
4. Any contraindication against the use of vagolytic or sympaticomimetic drugs, as judged by the Investigator.
5. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
6. Any clinically significant abnormalities in clinical chemistry, hematology, or urinalysis results, as judged by the Investigator.
7. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (anti HBc Ab), hepatitis C antibody and human immunodeficiency virus (HIV).
8. Abnormal vital signs, after 10 minutes supine rest (confirmed by 1 controlled measurement), defined as any of the following:

   * Systolic BP (SBP) < 90 mmHg or ≥ 140 mmHg
   * Diastolic BP (DBP) < 50 mmHg or ≥ 90 mmHg
   * Pulse < 50 or > 90 beats per minute (bpm)
9. Subject with forced expiratory volume in 1 second (FEV1) < 80% of the predicted value regarding age, height, gender and ethnicity (European Community for Coal and Steel [ECCS/European Respiratory Society [ERS]) at screening.
10. Subject with an acute infection of the upper and lower airway or other clinical relevant infections, which are not resolved at least 3 weeks before first drug administration.
11. Subjects who are not able to perform correct spirometry tests at screening.
12. Any clinically significant abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically significant abnormalities in the 12 lead ECG, as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST T wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy.
13. Prolonged Fridericia's correction (QTcF) > 450 ms or family history of long QT syndrome.
14. PR (PQ) interval prolongation (> 200 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.
15. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of, for example, ventricular hypertrophy or pre excitation.
16. Known or suspected history of drug abuse, as judged by the Investigator.
17. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the previous 3 months.
18. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
19. Positive screen for drugs of abuse or cotinine (nicotine) at screening or admission to the Clinical Unit.
20. History of severe allergy/hypersensitivity or ongoing clinically significant allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD7594.
21. Excessive intake of caffeine containing drinks or food (e.g., coffee, tea, chocolate), as judged by the Investigator.
22. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
23. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.
24. Plasma donation within one month of screening or any blood donation/blood loss > 500 mL during the 3 months prior to screening.
25. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest.

    Note: Subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
26. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.
27. Involvement of any Astra Zeneca or study site employee or their close relatives.
28. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
29. Subjects who are vegans or have medical dietary restrictions.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) of abediterol and AZD7594 from time zero extrapolated to infinity. AUC is estimated by AUClast + Clast/λz where Clast is the last observed quantifiable concentration | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Maximum observed plasma concentration (AUClast), taken directly from the individual concentration time curve of abediterol and AZD7594. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Observed maximum concentration (Cmax) of abediterol and AZD7594, taken directly from the individual concentration time curve. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) of abediterol and AZD7594 using plasma concentrations, estimated as (ln2)/λz. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Time to reach maximum observed plasma concentration (tmax) of abediterol and AZD7594 using plasma concentrations, taken directly from the individual concentration time curve. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Mean residence time (MRT) of abediterol and AZD7594. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Apparent estimated as dose divided by AUC.total body clearance of drug from plasma after extravascular administration (CL/F) of abediterol and AZD7594, | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
The time interval (h) of the log linear regression to determine t1/2λz (λz upper and λz lower) of abediterol and AZD7594. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Terminal elimination rate constant, estimated by log linear least squares regression of the terminal part of the concentration time curve (λz, N) of abediterol and AZD7594. | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Regression coefficient adjusted for λz, N observations, goodness of fit statistic for calculation of λz (Rsq_adj) of abediterol and AZD7594 | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs
Percentage of AUC obtained by extrapolating the area under the plasma concentration time curve from the time of the last quantifiable concentration to infinity (%AUCextr) of abediterol and AZD7594 | Day -1 to Day 3. Subjects will also return to the Unit at 72, 96, 144 and 240 hours post-dose (Days 4, 5, 7 and 11 respectively) for PK measurements
  Pharmacokinetics of AZD7594 and abediterol following single inhaled doses of AZD7594 alone, abediterol alone and the 2 compounds in FDC or in free combination via 2 separate DPIs

SECONDARY OUTCOMES:
Safety and tolerability of single inhaled doses of AZD7594 and abediterol alone and in combination assessed by recording the AEs, physical examination, electrocardiogram readings, vital signs, spirometry and clinical laboratory assessments. | From Screening (maximum of 28 days) till Follow up visit (10 to 14 days post final dose), an average of 24 weeks
  Safety and tolerability of single inhaled doses of AZD7594 and abediterol alone and in combination in healthy male subjects will be assessed by recording the AEs, physical examination, electrocardiogram (12-lead paper print-out ECG [pECG], digital ECG [dECG] and telemetry), vital signs (pulse rate, BP and oral body temperature), spirometry and clinical laboratory assessments (hematology, clinical chemistry including serum potassium and glucose and urinalysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Berlin, Germany